CLINICAL TRIAL: NCT04875546
Title: An Integrated Smoking Cessation and Alcohol Intervention Among Hong Kong Chinese Young People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Smk_AI-RCT
Record Dates: First submitted 2021-04-20; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Adolescent Behavior
Keywords: smoking; alcohol; adolescents
MeSH Terms: conditions — Adolescent Behavior; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment (Active Comparator): * A 5'A' and '5'R' models
  * STAR method for quitting
  Interventions: Behavioral: Standard treatment
- Integrated Intervention (Active Comparator): * A 5'A' and '5'R' models
  * Receive brief advice on alcohol use based on the FRAMES model
  * Complete the Alcohol Use Disorders Identification Test
  Interventions: Behavioral: Integrated Intervention
- Control (Sham Comparator): Participants will receive two leaflets.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Standard treatment — Adolescent will receive a brief smoking cessation intervention based on the '5A' and '5R' models. Then the research assistant will ask about their tobacco use and assist them to quit using the STAR method. A booster intervention will be given over the phone at 1-week, 1month, 3-month, and 6 month follow-up.
  Arms: Standard treatment
Behavioral: Integrated Intervention — In addition to the brief smoking cessation intervention based on the '5A' and '5R' models, the participants will receive brief advice on alcohol use based on the FRAMES model. Then the RA will invite participants to complete the Alcohol Use Disorders Identification Test and provide personalized feedback. There will be a one to one, 20-30 minutes semi-structured interviews with 30 participants. Participants with high(N=15) and low (N=15) adherence will be purposively selected. A booster intervention will be given over the phone at 1-week, 1month, 3-month, and 6 month follow-up.
  Arms: Integrated Intervention
Other: Control — The adolescents will receive the leaflets for smoking cessation and alcohol abstinence. A booster intervention will be given over the phone at 1-week, 1month, 3-month, and 6 month follow-up.
  Arms: Control

SUMMARY:
Current smoking cessation interventions are focused only on smoking behaviors, and drinking habits are generally overlooked. The aims of the project is to examine the feasibility of implementing an integrated smoking cessation and alcohol abstinence intervention in young Hong Kong Chinese smokers.

DETAILED DESCRIPTION:
The study is a three-arm randomized controlled trial. (1)The standard treatment group , participants will receive a brief smoking cessation intervention based on the '5A' and '5R' model, then the RA will assist the participants to quit smoking using the STAR method. (2) For the alcohol intervention group, participants will also receive a brief smoking cessation intervention with the models as the ST group. After that they will receive a brief advice on alcohol use based on the FRAMES model. Then the RA will invite participants to complete the Alcohol Use Disorders Identification Test(AUDIT). (3) For the Control group, participants will be provide with two leaflets, one for smoking cessation and another for alcohol abstinence. All the data collection will be conducted at baseline, 1 week, 1 month , 3 months and 6 months for follow up.

ELIGIBILITY:
Inclusion Criteria:

* smoked at least one cigarette in the past 30 days.
* have consumed at least one cup of alcohol in the past 30 days.
* speak Cantonese

Exclusion Criteria:

* have a compromised mental status and/or communication problems.
* participating in other smoking cessation interventions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The biochemical validation | At the 6-month follow-up
  Measuring the level of carbon monoxide in expired air and level of cotinine in saliva
Structured questionnaire | At baseline
  The questionnaire will include six areas: smoking profile, cessation history, readiness to quit, self-efficacy to quit, alcohol use and demographics.

SECONDARY OUTCOMES:
Randomization rate | Immediately after the training workshop
  The number of participants who randomized divided by the number of eligible smokers who consent to participate
Attendance rate | Immediately after the training workshop
  The number of participants who complete intervention divided by the number of participants who are randomized into the treatment arms participants who are randomized into the treatment arms
Adherence to intervention at baseline | At baseline
  The number of participants in the two treatment arms who practice the skills learned during the intervention divided by the number of participants in the two treatment arms during the intervention divided by the number of participants in the two treatment arm.
Adherence to intervention at 1-week follow-up | At 1-week follow-up
  The number of participants in the two treatment arms who practice the skills learned during the intervention divided by the number of participants in the two treatment arms during the intervention divided by the number of participants in the two treatment arm.
Adherence to intervention at 1-month follow-up | At 1-month follow-up
  The number of participants in the two treatment arms who practice the skills learned during the intervention divided by the number of participants in the two treatment arms during the intervention divided by the number of participants in the two treatment arm.
Adherence to intervention at 3-month follow-up | At 3-month follow-up
  The number of participants in the two treatment arms who practice the skills learned during the intervention divided by the number of participants in the two treatment arms during the intervention divided by the number of participants in the two treatment arm.
Adherence to intervention at 6-month follow-up | At 6-month follow-up
  The number of participants in the two treatment arms who practice the skills learned during the intervention divided by the number of participants in the two treatment arms during the intervention divided by the number of participants in the two treatment arm.
Retention rate at baseline | At baseline
  The number of participants who remain in the study divided by the number of participants randomized. Retention rate will be calculated for each arm at baseline and follow-ups.
Retention rate at 1-week follow-up | At 1-week follow-up
  The number of participants who remain in the study divided by the number of participants randomized. Retention rate will be calculated for each arm at baseline and follow-ups.
Retention rate at 1-month follow-up | At 1-month follow-up
  The number of participants who remain in the study divided by the number of participants randomized. Retention rate will be calculated for each arm at baseline and follow-ups.
Retention rate at 3-month follow-up | At 3-month follow-up
  The number of participants who remain in the study divided by the number of participants randomized. Retention rate will be calculated for each arm at baseline and follow-ups.
Retention rate at 6 month follow-up | At 6-month follow-up
  The number of participants who remain in the study divided by the number of participants randomized. Retention rate will be calculated for each arm at baseline and follow-ups.
Completion rate at baseline | At baseline
  The number of participants who complete the questionnaire divided by the number of questionnaires distributed.
Completion rate at 1-week follow-up | At 1-week follow-up
  The number of participants who complete the questionnaire divided by the number of questionnaires distributed.
Completion rate at 1-month follow-up | At 1-month follow-up
  The number of participants who complete the questionnaire divided by the number of questionnaires distributed.
Completion rate at 3-month follow-up | At 3-month follow-up
  The number of participants who complete the questionnaire divided by the number of questionnaires distributed.
Completion rate at 6-month follow-up | At 6-month follow-up
  The number of participants who complete the questionnaire divided by the number of questionnaires distributed.
Missing data at baseline | At baseline
  The percentage of missing data.
Missing data at 1-week follow-up | At 1-week follow-up
  The percentage of missing data.
Missing data at 1-month follow-up | At 1-month follow-up
  The percentage of missing data.
Missing data at 3-month follow-up | At 3-month follow-up
  The percentage of missing data.
Missing data at 6-month follow-up | At 6-month follow-up
  The percentage of missing data.
Adverse events | At the 6 months follow up
  Unfavorable or unintended events during the study period that were not present at baseline or appear to have worsened since baseline
Screen rate | Immediately after the training workshop
  The number of people screened divided by the number of people available for screening.
Consent rate | Immediately after the training workshop
  The number of eligible smokers who agree to participate divided by the number of eligible smokers
Eligibility rate | Immediately after the training workshop
  The number of eligible smokers divided by the number of screened people.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, Phd, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Ka Yan Ho, Hong Kong, Hong Kong,China, Hong Kong

IPD SHARING:
Plan to Share IPD: No